CLINICAL TRIAL: NCT02480465
Title: Efficacy and Safety of Lobeglitazone Versus Sitagliptin in Inadequately Controlled by Metformin Alone Type 2 Diabetes Mellitus Patients With Metabolic Syndrome: 24-week, Multi-center, Randomized, Double-blind, Phase 4 Study
Brief Title: Efficacy and Safety of Lobeglitazone Versus Sitagliptin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39DM14010
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lobelitazone 0.5mg (Experimental): Lobelitazone 0.5mg
  Interventions: Drug: Lobelitazone 0.5mg
- Sitagliptin 100mg (Active Comparator): Sitagliptin 100mg
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Lobelitazone 0.5mg — Lobelitazone 0.5mg, placebo of Sitagliptin 100mg, orally, 2 tablet once a day for 24 weeks with metformin
  Arms: Lobelitazone 0.5mg
Drug: Sitagliptin 100mg — placebo of Lobelitazone 0.5mg, Sitagliptin 100mg, orally, 2 tablet once a day for 24 weeks with metformin
  Arms: Sitagliptin 100mg

SUMMARY:
Efficacy and Safety of Lobeglitazone versus Sitagliptin in inadequately controlled by Metformin alone Type 2 Diabetes mellitus Patients with Metabolic syndrome.

DETAILED DESCRIPTION:
Efficacy and Safety of Lobeglitazone versus Sitagliptin in inadequately controlled by Metformin alone Type 2 Diabetes mellitus Patients with Metabolic syndrome: 24-week, Multi-center, Randomized, Double-blind, Phase 4 Study.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years old
* Waist line: male ≥ 90cm, female ≥ 85cm
* Applied to 1 or more categories listed below (NCEP-ATP III)

  1. SBP ≥ 130mmHg and/or DBP ≥ 85mmHg and/or taking drug for BP control
  2. HDL-C: male < 40mg/dl, female < 50mg/dl and/or taking drug for HDL-C increase
  3. TG ≥ 150mg/dl and/or taking drug for TG control
* At visit 1: Applied to 1 or more categories listed below

  1. Type 2 DM Patients who does not need stabilization period : 7% ≤ HbA1c ≤ 10%, if treated with Metformin ≥ 1000mg monotherapy at least 12 weeks prior to this study → Visit 3(Randomization)
  2. Type 2 DM Patients who need stabilization period : 7% ≤ HbA1c ≤ 10%, if not treated with Metformin ≥ 1000mg monotherapy at least 12 weeks prior to this study (Applied to 1 or more categories listed below) ① Drug Naïve ② Taking Metformin < 1000mg monotherapy and/or Taking Metformin < 12 weeks prior to this study ③ Taking OHA
* At visit 2(After 12 weeks of stabilization period): 7% ≤ HbA1c ≤ 10%
* Patients who signed informed consent form

Exclusion Criteria:

* Type 1 DM Patients or secondary DM
* Patients with ketoacidosis
* Patients with taking insulin > 7 days within 12 weeks
* Hypersensitive to biguanide and/or glitazone and/or DPP4-inhibitor
* Patients with taking corticosteroid > 7 days within 4 weeks
* Patients with lactic acidosis
* Patients with galactose intolerance and/or Lapp lactase deficiency and/or glucose-galactose malabsorption
* Patients with innutrition and/or starvation and/or weakness and/or pituitary insufficiency and/or addisons disease
* History of malignant tumor within 5 years
* History of drug or alcohol abuse within 12 weeks
* Patients with congestive heart failure(NYHA class III~IV) or uncontrolled arrythmia within 6 months
* Patients with acute cardiovasvular disaese with 12 weeks
* Applied to 1 or more categories listed below

  1. AST and/or ALT ≥ 3*ULN
  2. Serum creatinine: male ≥ 1.5mg/dl, female ≥ 1.4mg/dl
  3. Hb < 10.5g/dl
* Women with pregnant, breast-feeding
* Childbearing age who don't use adequate contraception
* Patients who have participated in other clinical trials
* Not eligible to participate for the study at the discretion of investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The mean percent change of HbA1c | from baseline at 24 weeks

SECONDARY OUTCOMES:
The rate of Metabolic Syndrome | from baseline at 24 weeks
The mean percent change of Metabolic Syndrome Components(HDL-C, TG, BP, waist line) | from baseline at 24 weeks
The mean percent change of Glycemic parameters(FPG, HOMA-IR, HOMA- β, QUICKI) | from baseline at 24 weeks
The mean percent change of Lipid parameters(Total Cholesterol, LDL-C, HDL-C, Small Dense LDL-C, FFA, Apo-B) | from baseline at 24 weeks
The achivement rate of HbA1c(HbA1c < 6.5%, HbA1c < 7%) | from baseline at 24 weeks
The mean percent change of Adiponectin | from baseline at 24 weeks
The mean percent change of hs-CRP | from baseline at 24 weeks
Safety evaluation - physical examination, vital sign, laboratory, adverse event | from baseline at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Sub Choi, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea